CLINICAL TRIAL: NCT03260816
Title: Advancing Child Competencies by Extending Supported Services (ACCESS) for Families Program
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of Miami (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-15-0134; R01HD084497 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Developmental Delay; Disruptive Behavior
Keywords: Preschoolers; Developmental Delay; Disruptive Behavior; Early Intervention; Parent-Child Interaction Therapy (PCIT); Telehealth; Telemental Health; Telepsychiatry
MeSH Terms: conditions — Learning Disabilities; Problem Behavior | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Randomized control trial in which participants are randomly assigned to either receive Internet-delivered Parent-Child Interaction Therapy (I-PCIT) or referrals as usual (RAU).
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators and coders assessing response over time are kept unaware of the condition to which each participant is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Delivered Parent Training (Experimental): Families will receive weekly sessions of Internet-delivered Parent-Child Interaction Therapy (I-PCIT), a short-term parent-training intervention emphasizing positive attention, consistency, problem-solving, and communication. Using videoconferencing, webcams, and wireless Bluetooth earpieces, I-PCIT therapists provide in-the-moment feedback to parents during live parent-child interactions.
  Interventions: Behavioral: Internet-delivered Parent-Child Interaction Therapy (I-PCIT)
- Referrals as Usual (RAU) (Active Comparator): Families in the referrals as usual (RAU) group will be referred to services as usual in their Early Intervention exit interview, which includes a variety of clinic-based mental health services at local community agencies. At each assessment, the access and extent of participation in other services will be monitored.
  Interventions: Other: Referrals as Usual (RAU)

INTERVENTIONS:
Behavioral: Internet-delivered Parent-Child Interaction Therapy (I-PCIT) — Families assigned to the Internet-delivered Parent-Child Interaction Therapy (I-PCIT) group will receive Internet-delivered weekly sessions of a short-term parent-training intervention emphasizing positive attention, consistency, problem-solving, and communication. Using videoconferencing, webcams, and wireless Bluetooth earpieces, I-PCIT therapists provide in-the-moment feedback to parents during live parent-child interactions.
  Arms: Internet-Delivered Parent Training
Other: Referrals as Usual (RAU) — Families assigned to RAU will participate in services referred by their Early Steps team, as per usual care.
  Arms: Referrals as Usual (RAU)

SUMMARY:
The Advancing Child Competencies by Extending Supported Services (ACCESS) for Families Program is a study funded by the National Institutes of Health to explore behavior and developmental problems among young children aging out of Early Steps (Part C). All families will participate in five evaluations in their home to learn more about their child's behavior and development. Families also may receive treatment designed to help change their child's behaviors that will be conducted over the Internet using a tablet.

DETAILED DESCRIPTION:
The proposed study will evaluate, via a randomized controlled trial, the incremental utility of I-PCIT for disruptive behavioral problems in traditionally underserved young children with developmental delay (DD) from predominantly economically disadvantaged and ethnic and racial minority backgrounds. Specifically, the investigators are interested in the impact of I-PCIT on child disruptive behavior problems, parenting practices, parental distress, and pre-academic skills relative to traditional referrals as usual (RAU) among youth aging out of Part C EI services and transitioning from home-based family services to school-based special education services. A secondary goal is to evaluate potential moderators and mediators that explain under which circumstances, for whom, and through which pathways I-PCIT is most effective for young children with DD. Our primary aims are (1) to evaluate the immediate and one-year impact of I-PCIT on (1a) disruptive behavior problems in young children with DD, as well as (1b) parenting practices and (1c) parental distress in parents of young children with DD; (2) to evaluate the impact of I-PCIT on pre-academic skills among young children with DD; and (3) to evaluate (3a) family retention, (3b) engagement, and (3c) satisfaction associated with I-PCIT in young children with DD. Our secondary aim is to examine potential moderators and mediators of response to I-PCIT for disruptive behavior problems in young children with DD. Specifically, the investigators are interested in the extent to which technological literacy and access (4a) moderate I-PCIT efficacy, such that I-PCIT efficacy will be weaker among families with poorer technological literacy and/or access, and the extent to which traditional barriers to care (4b) moderate I-PCIT efficacy, such that the incremental efficacy of I-PCIT over RAU will be strongest among families with geographic, transportation and/or childcare obstacles to in-person services. Finally, the investigators hypothesize that I-PCIT will yield changes in child behavior and pre-academic skills indirectly through direct effects on parenting practices (4c). Specifically, changes in parental consistency, warmth, follow-through, and effective discipline will mediate observed I-PCIT efficacy, such that these treatment-related parenting changes will account for observed differences in child disruptive behavior problems and pre-academic skills.

ELIGIBILITY:
Inclusion Criteria:

* Young children aging out of Part C EI services (mean age = 34.50 months) and at least 1 primary caretaker, which in most cases will be the mother
* Elevated Child Behavior Checklist Externalizing Problems scale at least in the borderline clinical range (i.e., T-score = 60)
* English-speaking or Spanish-speaking primary caretaker and child.

Exclusion Criteria:

* Child receiving an unstable dose of medication (i.e., changes within the past 4 weeks) to manage behavior difficulties
* History of severe physical impairment (e.g., deafness, blindness) in the child or primary caretaker
* Severe autism spectrum disorder impairment (i.e., Social Responsiveness Scale, Second Edition > 75)
* Significant cognitive delay in the parent (i.e., estimated IQ score < 70 on the two-subtest [vocabulary and matrix reasoning] version of the Wechsler Abbreviated Scale of Intelligence for those speaking English or an average standard score < 4 on the vocabulary and matrix reasoning subtests of the Escala de Inteligencia Wechsler Para Adultos - Third Edition for those speaking Spanish)

Ages: 30 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist, Ages 1.5-5 (CBCL, 1.5-5) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Child Behavior Checklist 1.5-5 (CBCL/1.5-5; Achenbach & Rescorla, 2001) is a 99-item caregiver- report questionnaire of behavioral, emotional, and social problems in children between the ages of 18 months and 5 years. In the current study the externalizing behavior problem scale will be used to screen children into the study (T- score = 60), and the following subscales will be used as outcomes: aggressive behavior, attention problems, attention-deficit/hyperactivity problems, emotionally reactive, and oppositional defiant problems.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline (Week 0), Post (Week 21), Follow-Up One (Week 42) and Follow-Up Two (Week 68)
  A weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters.
Sutter-Eyberg Behavior Inventory, Revised (SESBI-R) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R; Eyberg & Pincus, 1999) is a teacher rating scale of disruptive behaviors at school in children as young as 2 years, and the Intensity and Problem scales will be used as outcome measures for participants in school to assess generalization of improvement in child disruptive behavior to the classroom setting.
Multidimensional Assessment of Preschool Disruptive Behavior (MAP-DB): Temper Loss Scale | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Temper Loss Scale of the Multidimensional Assessment of Preschool Disruptive Behavior (MAP-DB; Wakschlag et al., 2014) assesses temper loss in terms of tantrum features and anger regulation.
Impossibly Perfect Circle (IPC) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  Children will complete a self-regulation task called the Impossibility Perfect Circles (IPC; Goldsmith & Reilly, 1993) task in which the child is asked to draw a perfect circle several times. The purpose of this task is to code how well the child is regulating their behaviors and emotions during challenging tasks.
Child Rearing Inventory (CRI) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Child Rearing Inventory (CRI; Brestan et al., 2003) is an 11-item caregiver-report measure of caregivers' ability to tolerate misbehavior and will also be used as an outcome measure of parenting practices.
Parenting Practices Inventory (PPI) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Parenting Practices Inventory (PPI; Webster-Stratton et al., 2004)) is a 72-item caregiver-report questionnaire designed to measure caregiver disciplinary styles and strategies. The PPI is designed to measure parenting practices using the following subscales: appropriate discipline, harsh and inconsistent discipline, positive verbal discipline, monitoring, physical punishment, praise and incentives, and clear expectations.
Parent-Child Book Reading | Change from Week 0, Week 21, Week 42 and Week 68
  The caregiver-child book- reading procedure will consist of one age-appropriate book (The Way I Feel by Janan Cain; Cain, 2005) which also has Spanish version (Asi me siento yo by Janan Cain; Cain, 2009). Caregivers will be instructed to describe the books to their children like they would normally for 5 minutes. This book is intended to elicit emotion talk as it includes emotional content, but also depicted multiple scenes, events, and objects that caregivers could talk about in addition to or instead of emotions, thereby permitting the capture of differences in caregivers' predilection to discuss emotions with their children.
Family Impact Questionnaire (FIQ) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Family Impact Questionnaire (FIQ; Donenberg & Baker, 1993) is a 50-item caregiver-report questionnaire of stress and strain, selected over other measures as an outcome of caregiver distress because it has been Child Disruptive Symptoms.
Depression, Anxiety, Stress Scale- 21 (DASS-21) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Depression, Anxiety, Stress Scale-21 (DASS21; Lovibond & Lovibond, 1995) is a clinical assessment that measures the three related states of depression, anxiety and stress.
Bracken School Readiness Assessment-3 (BSRA-3) | Change from Week 0, Week 21, Week 42 and Week 68
  Bracken School Readiness Assessment-3 (BSRA-3; Bracken, 2007) is an individual cognitive test designed for children examining the areas of colors, letters, numbers/counting, sizes, comparisons, and shapes.
Preschool Language Scale-5 (PLS-5) | Change from Week 0, Week 21, Week 42 and Week 68
  The Preschool Language Scale-5 (PLS-5; Zimmerman, Steiner, & Pond, 2011) is an assessment of developmental language skills, specifically auditory comprehension and expressive communication.
Clinical Global Impression (CGI-I) | Week 21
  The Clinical Global Impression - Improvement scale (CGI-I; Guy, 1976) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Technology Experience and Attitude Rating Scale (TEARS) | Change in weekly ratings from Week 0 to Week 21
  The Technology Experience and Attitude Rating Scale (TEARS) will be administered to assess caregiver and child technology use and literacy as a potential moderator of treatment response.
Therapy Attitude Inventory (TAI) | Week 21
  The Therapy Attitude Inventory (TAI; Brestan et al. 2000) is a 10-item parent-report of satisfaction with the process and outcome of parent-training interventions.
Client Satisfaction Questionnaire-8 (CSQ-8) | Week 21
  The Client Satisfaction Questionnaire-8 (CSQ-8; Nguyen et al., 1983) is an 8-item generic measure of clients' perceptions of the value of services received.
Telepresence in Videoconferencing Scale | Week 21
  The Telepresence in Videoconferencing Scale will be administered to assess caregiver experience interacting within video web-conferencing platform.
Barriers to Treatment Participation Scale (BTPS) | Week 21
  The Barriers to Treatment Participation Scale (BTPS; Kazdin et al. 1997) is a 44-item measure of perceived barriers to treatment participation.
Parental Attitudes Toward Psychological Services Inventory (PATPSI): Stigmatization Scale and Help-Seeking Attitudes Scale | Baseline (Week 0)
  Two scales from the Parental Attitudes Toward Psychological Services Inventory (PATPSI; Turner, 2012) will be administered: help- seeking attitudes scale and the stigmatization scale. The PATPSI is a measure to assess caregivers' attitudes toward outpatient mental health services.
Child's Sleep Habits Questionnaire | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Children's Sleep Habits Questionnaire (CSHQ; Owens et al. 2000) is a 33-item parent questionnaire designed to examine sleep behavior in young children and thus screen for the most common sleep problems.
Dyadic Parent-Child Interaction Coding System-IV (DPICS-4) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Dyadic Parent-Child Interaction Coding System-4th Ed (DPICS-IV; Eyberg et al., 2013) is a structured behavioral observation coding system assessing caregiver-child interactions. Observed parenting behaviors will be coded during a 5-min child-led play and combined into two categories of positive (praises, behavior descriptions, and reflections) and negative (questions, commands, and negative talk) verbalizations, reflecting behaviors caregivers are taught to use and avoid in PCIT. Additionally, child compliance will be assessed during a 5-min caregiver-led play and 5-min clean up situation and will be examined as an objective outcome of child behavior. The positive and negative caregiver verbalizations will be examined as both outcomes and candidate mediators of treatment, and child compliance will be examined as an outcome.
Eyberg Child Behavior Inventory (ECBI) | Change from Week 0, Week 8, Week 21, Week 42 and Week 68
  The Eyberg Child Behavior Inventory (ECBI; Eyberg & Pincus, 1999) is a 36-item caregiver-report of disruptive behavior problems in children as young as 2 years. The Intensity and Problem scales will be used to assess changes in child disruptive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Bagner, Ph.D., ABPP, Principal Investigator — Florida International University; Jonathan S. Comer, Ph.D., Principal Investigator — Florida International University
Locations (3):
- United States (3):
  - University of Miami, Early Steps North, Miami, Florida
  - Florida International University, Miami, Florida
  - Nicklaus Children's Hospital, Early Steps South, Palmetto Bay, Florida

IPD SHARING:
Plan to Share IPD: Undecided
We will use a controlled access approach, using a robust system to review requests and provide secure access to de-identified data.

REFERENCES:
- [Background] Achenbach, T. M., & Rescorla, L. A. (2001). Manual for the ASEBA Preschool Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Myers K, Cain S; Work Group on Quality Issues; American Academy of Child and Adolescent Psychiatry Staff. Practice parameter for telepsychiatry with children and adolescents. J Am Acad Child Adolesc Psychiatry. 2008 Dec;47(12):1468-83. doi: 10.1097/CHI.0b013e31818b4e13. PMID 19034191
- [Background] Bracken, B. A. (2007). Bracken School Readiness Assessment. San Antonio, TX: Psychological Corporation.
- [Background] Brestan , E. V. , Eyberg , S. M. , Algina , J. , Bennett Johnson , S. , & Boggs , S. R. ( 2003 ). How annoying is it? Defining parental tolerance for child misbehavior. Child and Family Behavior Therapy, 25, 1-15.
- [Background] Brestan, E. V., Jacobs, J. R., Rayfield, A. D., & Eyberg, S. M. (2000). A consumer satisfaction measure for parent-child treatments and its relation to measures of child behavior change. Behavior Therapy, 30, 17-30.
- [Background] Cain, J. (2005). The Way I Feel. Chicago, IL: Parenting Press.
- [Background] Cain, J. (2009). Asi Me Sientol. Chicago, IL: Parenting Press.
- [Background] Donenberg G, Baker BL. The impact of young children with externalizing behaviors on their families. J Abnorm Child Psychol. 1993 Apr;21(2):179-98. doi: 10.1007/BF00911315. PMID 8491931
- [Background] Eyberg, S. M., & Funderburk, B. W. (2011). Parent-Child Interaction Therapy Protocol. Gainesville, FL: PCIT International.
- [Background] Eyberg, S. M., Nelson, M. M., Ginn, N. C., Bhuiyan, N., & Boggs, S. R. (2013). Dyadic Parent- Child Interaction Coding System (DPICS): Comprehensive manual for research and training. Gainesville, FL: PCIT International.
- [Background] Eyberg, S. M., & Pincus, D. (1999). Eyberg Child Behavior Inventory and Sutter-Eyberg Student Behavior Inventory: Professional manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Goldsmith, H.H., Reilly, J (1993). Laboratory Assessment of Temperament Preschool Version. University of Oregon.
- [Background] Guy, W. (1976). ECDEU assessment manual for psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration.
- [Background] Hall, L. (1983). Social supports, everyday stressors, and maternal mental health (Unpublished doctoral dissertation). University of North Carolina at Chapel Hill.
- [Background] Jensen PS, Eaton Hoagwood K, Roper M, Arnold LE, Odbert C, Crowe M, Molina BS, Hechtman L, Hinshaw SP, Hoza B, Newcorn J, Swanson J, Wells K. The services for children and adolescents-parent interview: development and performance characteristics. J Am Acad Child Adolesc Psychiatry. 2004 Nov;43(11):1334-44. doi: 10.1097/01.chi.0000139557.16830.4e. PMID 15502592
- [Background] Kazdin AE, Holland L, Crowley M, Breton S. Barriers to Treatment Participation Scale: evaluation and validation in the context of child outpatient treatment. J Child Psychol Psychiatry. 1997 Nov;38(8):1051-62. doi: 10.1111/j.1469-7610.1997.tb01621.x. PMID 9413802
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety & Stress Scales. (2 Ed.)Sydney: Psychology Foundation.
- [Background] Newborg J. (2005). Battelle developmental inventory-second edition. Itasca, IL: Riverside.
- [Background] Newborg J. (2016) Battelle developmental inventory-second edition normative update. Itasca, IL: Riverside.
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Pons, J. I., Flores-Pabón, L., Matías-Carrelo, L., Rodríguez, M., Rosario-Hernández, E., Rodríguez, J. M., . . . Yang, J. (2008). Confiabilidad de la Escala de Inteligencia Wechsler para Adultos Versión III, Puerto Rico (EIWA-III). Revista Puertorriqueña de Psicología, 19, 112-132.
- [Background] Turner EA. The parental attitudes toward psychological services inventory: adaptation and development of an attitude scale. Community Ment Health J. 2012 Aug;48(4):436-49. doi: 10.1007/s10597-011-9432-7. Epub 2011 Jun 21. PMID 21691821
- [Background] Wakschlag LS, Briggs-Gowan MJ, Choi SW, Nichols SR, Kestler J, Burns JL, Carter AS, Henry D. Advancing a multidimensional, developmental spectrum approach to preschool disruptive behavior. J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):82-96.e3. doi: 10.1016/j.jaac.2013.10.011. Epub 2013 Nov 7. PMID 24342388
- [Background] Webster-Stratton C, Reid MJ, Hammond M. Treating children with early-onset conduct problems: intervention outcomes for parent, child, and teacher training. J Clin Child Adolesc Psychol. 2004 Mar;33(1):105-24. doi: 10.1207/S15374424JCCP3301_11. PMID 15028546
- [Background] Wechsler, D. (1999). Wechsler Abbreviated Scale of Intelligence. San Antonio, TX: Pychological Corportation.
- [Background] Zea MC, Asner-Self KK, Birman D, Buki LP. The abbreviated multidimensional acculturation scale: empirical validation with two Latino/Latina samples. Cultur Divers Ethnic Minor Psychol. 2003 May;9(2):107-126. doi: 10.1037/1099-9809.9.2.107. PMID 12760324
- [Background] Zimmerman, I.L., Steiner, V.G. and Pond, R.E., 2011, Preschool Language Scale, 5th Edition. (San Antonio, TX: The Psychological Corporation).
- [Derived] Cafatti Mac-Niven A, Comer JS, Bagner DM. Predictors of homework engagement in internet-delivered Parent-Child Interaction Therapy for children with developmental delay: what about acculturation and enculturation? Front Child Adolesc Psychiatry. 2025 Mar 12;4:1500742. doi: 10.3389/frcha.2025.1500742. eCollection 2025. PMID 40143964
- [Derived] Merrill SM, Hogan C, Bozack AK, Cardenas A, Comer JS, Bagner DM, Highlander A, Parent J. Telehealth Parenting Program and Salivary Epigenetic Biomarkers in Preschool Children With Developmental Delay: NIMHD Social Epigenomics Program. JAMA Netw Open. 2024 Jul 1;7(7):e2424815. doi: 10.1001/jamanetworkopen.2024.24815. PMID 39073812
- [Derived] Bagner DM, Berkovits MD, Coxe S, Frech N, Garcia D, Golik A, Heflin BH, Heymann P, Javadi N, Sanchez AL, Wilson MK, Comer JS. Telehealth Treatment of Behavior Problems in Young Children With Developmental Delay: A Randomized Clinical Trial. JAMA Pediatr. 2023 Mar 1;177(3):231-239. doi: 10.1001/jamapediatrics.2022.5204. PMID 36622653